CLINICAL TRIAL: NCT04677465
Title: A Clinical Evaluation of the RheOx Bronchial Rheoplasty System for the Treatment of the Symptoms of Chronic Bronchitis in Adult Patients With COPD
Brief Title: Clinical Study of the RheOx Bronchial Rheoplasty System in Treating the Symptoms of Chronic Bronchitis
Acronym: RheSolve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gala Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSP-00006
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-11

CONDITIONS: Chronic Bronchitis
Keywords: COPD
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Parallel group design randomizing patients in a 2:1 ratio to the treatment vs. sham group. Randomization will be blocked and stratified by site and FEV1 (<50% vs. >/= 50%)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RheOx Treatment (Experimental)
  Interventions: Device: RheOx Bronchial Rheoplasty
- Sham Procedure (Sham Comparator)
  Interventions: Device: Sham Procedure

INTERVENTIONS:
Device: RheOx Bronchial Rheoplasty — bronchial rheoplasty is a staged procedure wherein pulsed electric fields are delivered to the right lung in the first treatment visit, and then the left lung is treated approximately 1 month later.
  Arms: RheOx Treatment
Device: Sham Procedure — staged sham procedure wherein bronchoscopy is performed, the catheter is inserted into the right lung, but energy is not delivered; then the same steps are performed in the left lung approximately 1 month later (no energy is delivered to the patient)
  Arms: Sham Procedure

SUMMARY:
This is a prospective, randomized, parallel group, double-blind, sham-controlled, multicenter clinical trial following patients to 2 years. The objective is to assess the safety and effectiveness of Bronchial Rheoplasty for the treatment of the symptoms of chronic bronchitis in adult COPD patients with moderate to severe chronic bronchitis. A total of 270 patients will be randomized at up to 40 study centers in the United States, Canada, and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 35 years of age.
2. Patient has chronic bronchitis, defined as productive cough for three months in each of two successive years, whereas other causes of productive cough have been ruled out.
3. Patient has a CAT score ≥ 10.
4. Patient has an SGRQ score ≥ 25.
5. Patient's responses to the first two questions of the CAT instrument sum to ≥ 7 points or the sum is 6 points and the patient's total CAT score is > 20 points.
6. Patient has FEV1/FVC < 0.70.
7. Patient has a pre-procedure post-bronchodilator FEV1 percent predicted of ≥ 30%.
8. Patient is receiving guideline directed pharmacotherapy which includes one or more long acting bronchodilator (LAMA, LABA) with or without an inhaled corticosteroid for at least 8 weeks prior to randomization, unless the patient has attempted such therapy within the past 1 year without significant clinical response or had an adverse reaction.
9. Patient has a cigarette smoking history of at least ten pack years.
10. In the opinion of the Primary investigator, patient is able to undergo 2 bronchoscopies under general anesthesia and is able to adhere to the study follow-up schedule

Exclusion Criteria:

1. Patient has known unresolved lower respiratory tract infection (e.g., pneumonia, mycobacterium avium-intracellulare infection (MAI), fungus, tuberculosis).
2. Patient has a steroid-dependent condition requiring >10 mg of oral corticosteroid per day.
3. Patient has any implantable electronic device (e.g., pacemaker, cardioverter defibrillator) that cannot be turned off during the procedure.
4. Patient has a history of ventricular tachy-arrhythmia or clinically significant atrial tachyarrhythmia within the past two years, unless the arrhythmia has been treated and/or patient is in regular rhythm during the screening phase.
5. Patient has unresolved lung cancer.
6. Patient has a pulmonary nodule or cavity that in the judgement of the Primary investigator may require intervention during the course of the study.
7. Patient had prior lung surgery, such as lung transplant, LVRS, lobectomy, lung implant/prosthesis, metal airway stent, valves, coils or bullectomy. Prior pneumothorax without lung resection, pleural procedures without surgery, or segmentectomy are acceptable.
8. Patient has emphysema of greater than or equal to 25% as quantified on baseline HRCT scan (low attenuation area less than -950HU) as determined by the CT Core Lab.
9. Patient has asthma based on Global Initiative for Asthma (GINA) criteria.
10. Patient has clinically significant bronchiectasis influencing the patient's clinical symptoms of cough and phlegm.
11. Patient has actively smoked (including tobacco, marijuana, e-cigarettes, vaping, etc.) within the last 6 months.
12. Patient is unable to walk over 225 meters in 6 minutes.
13. Patient has a serious medical condition that, in the Primary investigator's opinion, could compromise patient safety or confound the interpretation of the patient's response to therapy (e.g., congestive heart failure, cardiomyopathy, or myocardial infarction in the past year, renal failure, liver disease cerebrovascular accident within the past 6 months, uncontrolled diabetes (HbA1c >8%), uncontrolled hypertension (diastolic BP >100mmHg) or autoimmune disease requiring treatment with immunosuppressant medications or a disease requiring chemotherapy).
14. Patient has uncontrolled GERD.
15. Patient has known severe pulmonary hypertension.
16. Patient has a known sensitivity to medication required to perform bronchoscopy (i.e., lidocaine, atropine, benzodiazepines).
17. Patient is pregnant, nursing, or planning to get pregnant during study duration.
18. Patient is currently participating in another clinical study involving an investigational product

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) Score | 6 months
  Mean change from baseline in the COPD Assessment Test (CAT) total score, the total CAT score ranges from 0 to 40, where lower scores represent lower symptom burden

SECONDARY OUTCOMES:
Distal Airway Volume | 6 months
  Change from baseline distal airway volume (DAV) at expiration using HRCT scans
COPD Exacerbations | 12 months
  Rate of moderate and severe COPD exacerbations
Goblet Cell Hyperplasia | 1 month
  change from baseline in mean goblet cell hyperplasia score as determined from airway biopsy samples; the grading scale ranges from 0 to 3, where lower scores represent less goblet cell hyperplasia
Cough Frequency | 6 and 12 months
  change from baseline in cough frequency (coughs/hour in a 24-hour recording period)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sciurba, MD, Principal Investigator — UPMC; Division of Pulmonary and Critical Care Medicine; Arschang Valipour, MD, Principal Investigator — Karl-Landsteiner-Institute for Lung Research and Pulmonary Oncology; Vienna, Austria
Locations (37):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Norton Thoracic, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - Syed M. Alam, MD Pulmonology (Bakersfield Heart), Bakersfield, California
  - UC Davis Medical Center, Davis, California
  - Scripps Health, Encinitas, California
  - University of Southern California, Los Angeles, California
  - UCLA Harbor Lundquist Institute, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - The Cardiac and Vascular Institute Research Foundation, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas School of Medicine, Kansas City, Kansas
  - Tulane University Medical Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - CHI Memorial Research Center, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - JPS Health Network, Fort Worth, Fort Worth, Texas
  - Houston Methodist, Houston, Texas
  - Virginia Commonwealth University Health, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Klinik Floridsdorf - Abteilung für Innere Medizin und Pneumologie, Vienna, Austria
- Germany (3):
  - Charité Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Ruhrlandklinik Essen, Essen
  - Thoraxklinik Heidelberg, Heidelberg
- ASST Spedali Civili Hospital, Brescia, Italy
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krimsky WS, VanderLaan PA, Iding JS, Hunter DW, Hatton BA, Bannan B, Kim V. A quantitative method for assessing treatment-related changes within the airway mucosa in patients with chronic bronchitis. Respir Med. 2025 Jan;236:107889. doi: 10.1016/j.rmed.2024.107889. Epub 2024 Nov 28. PMID 39615802